CLINICAL TRIAL: NCT04696315
Title: Comparison of Subjective Cognitive Decline Between the German and Chinese and Early Diagnosis of Alzheimer's Disease Based on Radiogenomics
Brief Title: Early Diagnosis of SCD Based on Radiogenomics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: XuanwuH 2 (Other)
Collaborators: University of Cologne (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: HanYingsc5
Record Dates: First submitted 2021-01-03; First posted 2021-01-06 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Alzheimer Disease; Subjective Cognitive Decline; Neuroimaging; Gene
Keywords: Subjective Cognitive Decline; Radiogenomics
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — In this project, the investigators will test ApoE, TREM2, p.P522R genotype.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCD subjects with positive amyloid: In this study, the participants are from two research centers in China and Germany. All participants will conduct amyloid PET scanning, after which they are classified into two grous (SCD with amyloid+ and SCD with amyloid-). SCD subjects with positive amyloid show the evidence of amyloid deposition in brain. They have higher risk of conversion to mild cognitive impairment and dementia compared with SCD with negative amyloid. They are also considered as preclinical AD.
  Interventions: Diagnostic Test: Multiple features extraction
- SCD subjects with negative amyloid: In this study, the participants are from two research centers in China and Germany. All participants will conduct amyloid PET scanning, after which they are classified into two grous (SCD with amyloid+ and SCD with amyloid-). SCD subjects with negative amyloid do not show the evidence of amyloid deposition in brain. They have lower risk of conversion to mild cognitive impairment and dementia compared with SCD with positive amyloid.
  Interventions: Diagnostic Test: Multiple features extraction

INTERVENTIONS:
Diagnostic Test: Multiple features extraction — In the present study, the "gold standard" of preclinical AD is amyloid PET. SCD with positive amyloid is the target population for early AD intervention. The investigators aim to extract the diagnostic features from multiple parameter MRI, genetic, blood and clinical data using Max-Relevance and Min-Redundancy (mRMR) algorithm. Then, based on support vector machine (SVM), random forest (RF) and multi-kernel learning (MKL) classification methods, the investigators will construct predicted diagnostic model of preclinical AD.

SUMMARY:
The incidence of AD dementia is increasing due to the aging population, putting a heavy burden on our society and economics. Exploring the mechanisms underlying SCD due to preclinical AD has scientific and clinical significance. However, it is challenging to construct and validate the preclinical diagnosis model of AD with fused multimodel information across culture/race. From the cooperation during the past five years, we have established cohorts by synchronized assessment, achieved consensus on SCD features extraction and made a breakthrough in the application of multiple parameter MRI with German collaborators. Therefore, in this project, SCD with and without amyloid pathology will be compared by clinical and cognitive data, genetics, blood and MRI biomarkers between the German and Chinese. Key features will be extracted and specific characteristics of SCD due to preclinical AD as well as risk factors for conversion between two countries will be clarified. Then the diagnosis model of preclinical AD in SCD will be established across culture/race based on radiogenomics, which will improve the current diagnostic system of AD. Through this project, the value of SCD in the etiologic, anatomical and quantitative diagnosis of preclinical AD will be identified to improve sensitivity and specificity of preclinical AD diagnosis in clinical practice.

DETAILED DESCRIPTION:
The overall prevalence of dementia worldwide is increasing, imposing a heavy burden on the public and health care systems. Subjective cognitive decline (SCD), characterized by a self-report of decline in cognitive function without objective impairment in neuropsychological assessments, is considered a high risk factor for AD. SCD with amyloidopathy is considered as a first symptomatic indicator of the preclinical AD (SCD due to preclinical AD). However, how to construct and validate the preclinical diagnosis model of AD with fused multimodel information across culture/race remain unclear.

In the present study, all SCD participants from Germany and China will be conducted amyloid PET scanning, and they will be classified into two groups (SCD with amyloid+ and SCD with amyloid-) based on whether there is the evidence of amyloid deposition. The investigators will compare the clinical information, genetics, blood and multiple parameter MRI data between the German and Chinese to evaluate the common and specific features from different culture/race. Then, key features associated with amyloid deposition will be extracted for the establisment of diagnosis model of SCD due to preclinical AD, which will improve the current diagnostic system of AD. After four-year follow-up, SCD will be classified into SCD converter group and SCD non-converter group. Risk factors for conversion to cognitive impairment and dementia will be further extracted as predicted biomarkers.

Through this project, the value of SCD in the etiologic, anatomical and quantitative diagnosis of preclinical AD will be identified to improve sensitivity and specificity of preclinical AD diagnosis in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 60-79 years old, right-handed and Mandarin-speaking subjects;
* self-experienced persistent decline in cognitive capacity in comparison with a previously normal status and unrelated to an acute event;
* normal age-, gender- and education-adjusted performance on standardised cognitive tests;
* concerns (worries) associated with memory complaint;
* failure to meet the criteria for MCI or dementia

Exclusion Criteria:

* a history of stroke;
* major depression (Hamilton Depression Rating Scale score > 24 points);
* other central nervous system diseases that may cause cognitive impairment, such as Parkinson's disease, tumors, encephalitis and epilepsy;
* cognitive impairment caused by traumatic brain injury;
* systemic diseases, such as thyroid dysfunction, syphilis and HIV;
* a history of psychosis or congenital mental growth retardation

Ages: 60 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: SCD may serve as a first symptomatic indicator during the preclinical stage of AD. SCD with amyloidopathy had a risk of progressing to AD dementia. In this study, all participants from two centers in Germany and China will be classified into two groups (SCD with amyloid+ and SCD with amyloid-) based on the amyloid PET. In addition, the participants will conduct multiple parameter MRI scanning, clinical data collection, blood biomarkers and gene examination. The investigators aim to reveal the common risk factors associated with amyloid deposition based on clinical, neuroimaging, and genetic information from two countries.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers associated with amyloid deposition | Four years
  SCD with the evidence of brain amyloid deposition is considered as preclinical AD. The investigators aim to extract multiple features involving neuroimaging, gene sequencing, blood, and clinical data to identify individuals with amyloid+ from SCD persons. These features associated with amyloid deposition are valuable biomarkers for early diagnosis of AD.

SECONDARY OUTCOMES:
Predicted biomarkers associated with conversion to cognitive impairment | Four years
  Individuals with SCD will be followed for four years. The investigators aim to characterize those who convert to mild cognitive impairment or dementia during the follow-up, and further find the predicted factors associated with the progression of AD.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University; Jessen Frank, PhD, Principal Investigator — University of Cologne
Locations (1):
- Department of Neurolgy, Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The information of neuropsychological tests, neuroimaging data are to be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: When summary data are published or starting 6 months after publication.
Access Criteria: The information of neuropsychological tests, neuroimaging data will be shared.

REFERENCES:
- [Derived] Shao K, Hu X, Kleineidam L, Stark M, Altenstein S, Amthauer H, Boecker H, Buchert R, Buerger K, Butryn M, Cai Y, Cai Y, Cosma NC, Chen G, Chen Z, Daamen M, Drzezga A, Duzel E, Essler M, Ewers M, Fliessbach K, Gaertner FC, Glanz W, Guo T, Hansen N, He B, Janowitz D, Kilimann I, Krause BJ, Lan G, Lange C, Laske C, Li Y, Li R, Liu L, Lu J, Meng F, Munk MH, Peters O, Perneczky R, Priller J, Ramirez A, Rauchmann BS, Reimold M, Rominger A, Rostamzadeh A, Roy-Kluth N, Schneider A, Spottke A, Spruth EJ, Sun P, Teipel S, Wang X, Wei M, Wei Y, Wiltfang J, Yan S, Yang J, Yu X, Zhang M, Zhang L; DELCODE study group, SILCODE study group; Wagner M, Jessen F, Han Y, Kuhn E. Amyloid and SCD jointly predict cognitive decline across Chinese and German cohorts. Alzheimers Dement. 2024 Sep;20(9):5926-5939. doi: 10.1002/alz.14119. Epub 2024 Jul 27. PMID 39072956
- [Derived] Sheng C, Yang K, He B, Li T, Wang X, Du W, Hu X, Jiang J, Jiang X, Jessen F, Han Y. Cross-Cultural Longitudinal Study on Cognitive Decline (CLoCODE) for Subjective Cognitive Decline in China and Germany: A Protocol for Study Design. J Alzheimers Dis. 2022;87(3):1319-1333. doi: 10.3233/JAD-215452. PMID 35431240